CLINICAL TRIAL: NCT05433896
Title: An Open Label, Non-Randomized, Two-Treatment, Single-Period, Single-Dose, Drug-Drug Interaction Study to Evaluate the Effects of Omeprazole on the Pharmacokinetics of XS004 (Dasatinib) 90 mg Film-Coated Tablets in Healthy Adult Subjects Under Fasting Conditions
Brief Title: Evaluating the Effects of Omeprazole on the Pharmacokinetics of XS004 (Dasatinib) Tablets in Healthy Adult Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xspray Pharma AB (Industry)
Collaborators: Axis Clinicals Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: XS004-09
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Pharmacokinetics; Drug Interactions
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dasatinib ASD alone (Experimental): At the clinic, participants were administered a single oral dose of 90 mg Dasatinib (Amorphous Solid Dispersion Film-Coated Tablet) on Day 1 after an overnight fast of at least 9 hours. Dasatinib was given with approximately 240 mL of room temperature water. Fasting continued for at least 4 hours following drug administration, after which a standardized lunch was served.
  Interventions: Drug: Dasatinib ASD
- Dasatinib ASD + Omeprazole (Other): At the clinic, on Day 2 to Day 6, participants were administered a single oral dose of Omeprazole 40 mg × 1 Delayed Release Capsule once before meals in the evening with approximately 150 mL of room temperature water. No food was allowed two hours before and one hour after administration of Omeprazole.
  In addition, participants were administered a single oral dose of 90 mg Dasatinib (Amorphous Solid Dispersion Film-Coated Tablet) on Day 6 after an overnight fast of at least 9 hours. Dasatinib was given with approximately 240 mL of room temperature water. Fasting continued for at least 4 hours following drug administration, after which a standardized lunch was served.
  Interventions: Drug: Dasatinib ASD; Drug: Omeprazole 40 MG

INTERVENTIONS:
Drug: Dasatinib ASD — XS004 Dasatinib Amorphous Solid Dispersion Film-Coated Tablet, 90 mg Test Formulation
Drug: Omeprazole 40 MG — Omeprazole Delayed Release Capsules, USP 40 mg
  Arms: Dasatinib ASD + Omeprazole

SUMMARY:
In this open label, single-sequence study, subjects received one dose of XS004 Dasatinib Amorphous Solid Dispersion Film-Coated Tablet, 90 mg Test Formulation at the start of study on Day 1 and Day 6. Omeprazole 40 mg was administered on Day 2, 3, 4, 5 and 6. The study was conducted in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* Sex: Healthy adult males (sterile or using contraception) and females of non-childbearing potential
* Clinical laboratory values should be within the laboratory's stated normal range. If not within this range, they must be without clinical significance, as determined by the Investigator
* No clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by the Investigator
* Any abnormalities/deviations from the acceptable range of medical history, laboratory values, ECG, and vital signs that might be considered clinically relevant by the study physician or Investigator will be evaluated as individual cases
* Able to comply with study procedures, in the opinion of the Investigator(s)
* Willing to give written consent, pregnancy outcome consent, and adhere to all the requirements of this protocol

Exclusion Criteria:

* Any major illness in the last three months or any significant ongoing chronic medical illness
* Does not agree to consume the provided meals
* Participation in any clinical trial 30 days prior to dosing
* Positive results for drugs of abuse or alcohol breath analysis prior to dosing
* Positive screening results to HIV Ag/Ab Combo, Hepatitis B surface Antigen, Hepatitis C Virus, or anti-HBc tests
* Females currently breastfeeding, demonstrating a positive pregnancy screen, or using hormone replacement therapy within three months prior to dosing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration of Dasatinib (Cmax) | Blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 6.
  Pharmacokinetic parameters (Cmax) for plasma dasatinib on Day 1 (Dasatinib alone) and on Day 6 (Dasatinib + Omeprazole) calculated for each subject using drug concentration-time data by non-compartmental methods.
Area Under the Plasma Concentration-Time Curve from Zero to 24h | Blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 6.
  Pharmacokinetic parameters (AUC 0-24) for plasma dasatinib on Day 1 (Dasatinib alone) and on Day 6 (Dasatinib + Omeprazole) calculated for each subject using drug concentration-time data by non-compartmental methods.
Area Under the Plasma Concentration-Time Curve from Zero Extrapolated to Infinity | Blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 6.
  Pharmacokinetic parameters (AUC 0-INF) for plasma dasatinib on Day 1 (Dasatinib alone) and on Day 6 (Dasatinib + Omeprazole) calculated for each subject using drug concentration-time data by non-compartmental methods.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve (Percent Extrapolation) | Blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 6.
  Pharmacokinetic parameters (AUC %Extrapolation) for plasma dasatinib on Day 1 (Dasatinib alone) and on Day 6 (Dasatinib + Omeprazole) calculated for each subject using drug concentration-time data by non-compartmental methods.
Time of Maximum Observed Plasma Concentration of Dasatinib (Tmax) | Blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 6.
  Pharmacokinetic parameters (Tmax) for plasma dasatinib on Day 1 (Dasatinib alone) and on Day 6 (Dasatinib + Omeprazole) calculated for each subject using drug concentration-time data by non-compartmental methods.
Elimination Rate Constant (Kel) | Blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 6.
  Pharmacokinetic parameters (Kel) for plasma dasatinib on Day 1 (Dasatinib alone) and on Day 6 (Dasatinib + Omeprazole) calculated for each subject using drug concentration-time data by non-compartmental methods. Apparent first order elimination rate constant calculated from a semi-log plot of plasma concentration versus time point.
Terminal Half-Life (T1/2) | Blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 6.
  Pharmacokinetic parameters (T1/2) for plasma dasatinib on Day 1 (Dasatinib alone) and on Day 6 (Dasatinib + Omeprazole) calculated for each subject using drug concentration-time data by non-compartmental methods.

CONTACTS AND LOCATIONS:
Overall Officials: Per Andersson, PhD, Study Director — Xspray Pharma AB
Locations (1):
- AXIS Clinicals, Dilworth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No